CLINICAL TRIAL: NCT03739710
Title: A Phase II, Randomized, Open-label Platform Trial Utilizing a Master Protocol to Study Novel Regimens Versus Standard of Care Treatment in NSCLC Participants
Brief Title: Platform Trial of Novel Regimens Versus Standard of Care (SoC) in Participants With Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: iTeos Belgium SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205801; 2018-001316-29 (EudraCT Number)
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms
Keywords: Non-small cell lung cancer; Inducible t-cell co-stimulator (ICOS); Docetaxel; Standard of care; Immuno-oncology agents; TIGIT; Dostarlimab; Jemperli; GSK4428859A; belrestotug; EOS884448; GSK6097608; Anti-TIGIT; CD-96; Anti-CD-96
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Ipilimumab; dostarlimab

STUDY DESIGN:
Masking Description: The study will be open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Participants receiving feladilimab and ipilimumab (Experimental)
  Interventions: Drug: Feladilimab; Drug: Ipilimumab
- Part 1: Participants receiving dostarlimab plus GSK4428859A/EOS884448/belrestotug (Experimental)
  Interventions: Drug: GSK4428859A; Drug: Dostarlimab
- Part 1: Participants receiving dostarlimab plus GSK4428859A/EOS884448/belrestotug plus GSK6097608 (Experimental)
  Interventions: Drug: GSK4428859A; Drug: Dostarlimab; Drug: GSK6097608
- Part 2: Participants receiving SoC: docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel
- Part 2: Participants receiving feladilimab and docetaxel (Experimental)
  Interventions: Drug: Docetaxel; Drug: Feladilimab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel will be administered.
  Arms: Part 2: Participants receiving SoC: docetaxel; Part 2: Participants receiving feladilimab and docetaxel
Drug: Feladilimab — Feladilimab will be administered.
  Arms: Part 1: Participants receiving feladilimab and ipilimumab; Part 2: Participants receiving feladilimab and docetaxel
Drug: Ipilimumab — Ipilimumab will be administered.
  Arms: Part 1: Participants receiving feladilimab and ipilimumab
Drug: GSK4428859A — GSK4428859A/EOS884448 will be administered.
  Other Names: belrestotug; EOS884448
  Arms: Part 1: Participants receiving dostarlimab plus GSK4428859A/EOS884448/belrestotug; Part 1: Participants receiving dostarlimab plus GSK4428859A/EOS884448/belrestotug plus GSK6097608
Drug: Dostarlimab — Dostarlimab will be administered.
  Arms: Part 1: Participants receiving dostarlimab plus GSK4428859A/EOS884448/belrestotug; Part 1: Participants receiving dostarlimab plus GSK4428859A/EOS884448/belrestotug plus GSK6097608
Drug: GSK6097608 — GSK6097608 will be administered.
  Arms: Part 1: Participants receiving dostarlimab plus GSK4428859A/EOS884448/belrestotug plus GSK6097608

SUMMARY:
This study will compare the clinical activity of novel regimens (in combination or as single agents) to SoC in participants with relapsed/refractory advanced NSCLC. The study will be conducted in two parts. Part 1 is an open-label, optional, non-randomized part based on safety and pharmacokinetics/pharmacodynamics (PK/PD) evaluation intended to generate additional data to qualify novel regimens for the randomized study. Part 2 is a randomized, Phase II open-label part comparing the efficacy and safety of these novel regimens with SoC. Drug name mentioned as GSK4428859A (belrestotug) and EOS884448 are interchangeable for the same compound and will be referred to as GSK4428859A/EOS884448/belrestotug.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of giving signed informed consent/assent.
* Male or female, aged 18 years or older at the time consent is obtained. Participants in Korea must be age 19 years or older at the time consent is obtained.
* Participants with histologically or cytologically confirmed diagnosis of NSCLC (squamous or non-squamous) and

  a) Documented disease progression based on radiographic imaging, during or after a maximum of 2 lines of systemic treatment for locally/regionally advanced recurrent, Stage IIIb/Stage IIIc/Stage IV or metastatic disease. Two components of treatment must have been received in the same line or as separate lines of therapy: i) No more than or less than 1 line of platinum-containing chemotherapy regimen, and ii) No more than or less than 1 line of Programmed cell death ligand 1 (PD[L]1) monoclonal antibody (mAb) containing regimen.

  b) Participants with known BRAF molecular alterations must have had disease progression after receiving the locally available SoC treatment for the molecular alteration.

  c) Participants who received prior anti-PD(L)1 therapy must fulfill the following requirements: i) Have achieved a CR, PR or SD and subsequently had disease progression (per RECIST 1.1 criteria) either on or after completing PD(L)1 therapy ii) Have not progressed or recurred within the first 12 weeks of PD(L)1 therapy, either clinically or per RECIST 1.1 criteria
* Measurable disease, presenting with at least 1 measurable lesion per RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
* A tumor tissue sample obtained at any time from the initial diagnosis of NSCLC to time of study entry is mandatory. Although a fresh tumor tissue sample obtained during screening is preferred, archival tumor specimen is acceptable.
* Adequate organ function as defined in the protocol.
* A male participant must agree to use a highly effective contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions apply:

  i) Not a woman of childbearing potential (WOCBP) or ii) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
* Life expectancy of at least 12 weeks.

Exclusion Criteria:

* Participants who received prior treatment with the following therapies (calculation is based on date of last therapy to date of first dose of study treatment):

  1. Docetaxel at any time.
  2. Any of the investigational agents being tested in the current study.
  3. Systemic approved or investigational anticancer therapy within 30 days or 5 half-lives of the drug, whichever is shorter. At least 14 days must have elapsed between the last dose of prior anticancer agent and the first dose of study drug is administered.
  4. Prior radiation therapy: permissible if at least one non-irradiated measurable lesion is available for assessment per RECIST version 1.1 or if a solitary measurable lesion was irradiated, objective progression is documented. A wash out of at least 2 weeks before start of study drug for radiation of any intended use is required.
* Received greater than (>)2 prior lines of therapy for NSCLC, including participants with BRAF molecular alternations.
* Invasive malignancy or history of invasive malignancy other than disease under study within the last 2 years, except

  * Any other invasive malignancy for which the participant was definitively treated, has been disease-free for at least 2 years and in the opinion of the principal investigator and GlaxoSmithKline Medical Monitor will not affect the evaluation of the effects of the study treatment on the currently targeted malignancy, may be included in this clinical trial.
  * Curatively treated non-melanoma skin cancer or successfully treated in situ carcinoma.
* Carcinomatous meningitis (regardless of clinical status) and uncontrolled or symptomatic Central nervous system (CNS) metastases.
* Major surgery less than or equal to (<=) 28 days of first dose of study treatment.
* Autoimmune disease (current or history) or syndrome that required systemic treatment within the past 2 years. Replacement therapies which include physiological doses of corticosteroids for treatment of endocrinopathies (for example, adrenal insufficiency) are not considered systemic treatments.
* Receiving systemic steroids (>10 milligrams [mg]) oral prednisone or equivalent) or other immunosuppressive agents within 7 days prior to first dose of study treatment.
* Prior allogeneic/autologous bone marrow or solid organ transplantation.
* Receipt of any live vaccine within 30 days prior to first dose of study treatment.
* Toxicity from previous anticancer treatment that includes:

  1. Greater than or equal to (>=) Grade 3 toxicity considered related to prior immunotherapy and that led to treatment discontinuation.
  2. History of myocarditis of any grade during a previous treatment with immunotherapy
  3. Toxicity related to prior treatment that has not resolved to <= Grade 1 (except alopecia, hearing loss, endocrinopathy managed with replacement therapy, and peripheral neuropathy which must be <= Grade 2).
* History (current and past) of idiopathic pulmonary fibrosis, pneumonitis (for past- pneumonitis exclusion only if steroids were required for treatment), interstitial lung disease, or organizing pneumonia.
* Recent history (within the past 6 months) of uncontrolled symptomatic ascites, pleural or pericardial effusions.
* Recent history (within the past 6 months) of gastrointestinal obstruction that required surgery, acute diverticulitis, inflammatory bowel disease, or intra-abdominal abscess.
* History or evidence of cardiac abnormalities within the 6 months prior to enrollment which include

  1. Serious, uncontrolled cardiac arrhythmia or clinically significant electrocardiogram abnormalities including second degree (Type II) or third degree atrioventricular block.
  2. Cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting or bypass grafting.
  3. Symptomatic pericarditis.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypo-albuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Active infection requiring systemic therapy <=7 days prior to first dose of study treatment.
* Participants with known human immunodeficiency virus infection.
* Participants with history of severe hypersensitivity to mAb or hypersensitivity to any of the study treatment(s) or their excipients.
* Participants requiring ongoing therapy with a medication that is a strong inhibitor or inducer of the cytochrome P 3A4 (CYP3A4) enzymes.
* Any serious and/or unstable pre-existing medical (aside from malignancy), psychiatric disorder, or other condition that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures in the opinion of the investigator.
* Pregnant or lactating female participants.
* Participant who is currently participating in or has participated in a study of an investigational device within 4 weeks prior to the first dose of study treatment.
* Participants with presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention.
* Participants with positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Participants with positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* Receipt of transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor, and recombinant erythropoietin) within 14 days before the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (52):
- United States (7):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Pinehurst, North Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Toronto, Ontario
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Villejuif
- Germany (7):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Gauting
  - GSK Investigational Site, Großhansdorf
  - GSK Investigational Site, Heidelberg
  - GSK Investigational Site, Immenhausen
  - GSK Investigational Site, Kassel
  - GSK Investigational Site, Leipzig
- Italy (6):
  - GSK Investigational Site, Meldola FC
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Orbassano to
  - GSK Investigational Site, Ravenna
  - GSK Investigational Site, Siena
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Maastricht
- Poland (3):
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- Romania (5):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Floreşti
  - GSK Investigational Site, Otopeni
  - GSK Investigational Site, Timișoara
- Russia (2):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Saint Petersburg
- South Korea (4):
  - GSK Investigational Site, Cheongju Chungcheongbuk-do
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, Badajoz
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
- Sweden (2):
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This master record includes data of screened participants for its sub-studies, 205801-001 (NCT05553808), 205801-002 (NCT06790303) and 205801-003 (NCT06926673) and only contains data during screening phase (Day -28 to Day 0). Results are presented separately for each sub study.
Pre-assignment Details: A total of 256 participants started the overall study which includes all who were screened prior to enrollment. However, 175 participants were enrolled in the study.
Groups:
- All Screened Participants: Participants with Non-Small Cell Lung Cancer (NSCLC) were screened to be enrolled in sub-studies of this master protocol.
Period: Overall Study
Arm/Group | All Screened Participants
Started (All participants who were screened for eligibility.) | 256
Completed (Enrolled in sub-studies) | 175
Not Completed | 81
Not completed — Screen Failed | 81

BASELINE CHARACTERISTICS:
Arm/Group | All Screened Participants
Number analyzed (Participants) | 256
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 127
  Over 64 years | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 170
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race categories ('Asian', 'Black or African American' and 'Native Hawaiian or Other Pacific Islander' where 0<n<11) are combined into 'All other races' category to maintain participant confidentiality and privacy.
  Participants
    White | 216
    Unknown or Not Reported | 12
    All other races | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Randomized Across Sub-studies
Description: Number of Participants randomized across sub studies are presented.
Time Frame: Day 1
Population: Randomized Population included all participants who passed screening and were assigned treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | All Screened Participants
Number analyzed (Participants) | 175
Participants
  Sub Study 1 | 105
  Sub Study 2 | 8
  Sub Study 3 | 62

ADVERSE EVENTS:
Time Frame: Screening (-28 to 0 days)
Description: Adverse event(s) of special interest [AESIs] and Serious Adverse Event(s) [SAEs] assessed as related to study participation, were not reported during the screening phase
Arm/Group | All Screened Participants
All-Cause Mortality (participants affected / at risk) | 0/256
Serious Adverse Events (participants affected / at risk) | 0/256
Other Adverse Events (participants affected / at risk) | 0/256

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT03739710/Prot_SAP_001.pdf